CLINICAL TRIAL: NCT04327973
Title: Expanded Use Of Recombinant Human Acid Alpha-Glucosidase/N-butyl-deoxynojirimycin (ATB200/AT2221) For Patients With Infantile-Onset Pompe Disease
Brief Title: Expanded Access for ATB200/AT2221 for the Treatment of IOPD
Status: Available | Type: Expanded Access
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: ATB200-15
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Pompe Disease Infantile-Onset
Keywords: expanded access; compassionate use

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: ATB200 — Participants received ATB200 co-administered with AT2221 capsule (Miglustat)
Drug: AT2221 — Participants received ATB200 co-administered with AT2221 capsule (Miglustat)

SUMMARY:
This is an expanded access program (EAP) for eligible participants designed to provide access to ATB200/AT2221.

DETAILED DESCRIPTION:
This program is being offered on a patient by patient basis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male or female and 0 to < 18 years old.
2. Patient has a diagnosis of Pompe disease, based on documentation of GAA genotyping demonstrating variants associated with IOPD.
3. Patient does not currently qualify for or is unable to enroll (eg, due to location, etc) in any commercial drug-sponsored ongoing clinical trial.
4. Patient is currently being treated with an approved ERT and is declining (eg, worsening in motor function, respiratory function/parameters, cardiac function, etc) based on treating physician's clinical judgement.
5. The patient's legal guardian or representative has given informed consent (and assent when age appropriate for regional requirements) to treatment prior to administering ATB200/AT2221 in a manner consistent with all national requirements.
6. If of reproductive potential and sexually active, female subjects agree to use a highly effective method of contraception throughout the duration of the treatment and for up to 90 days after their last dose of ATB200/AT2221.

Exclusion Criteria:

1. Patient has a hypersensitivity to any of the excipients in ATB200, alglucosidase alfa, or AT2221
2. Patient has a medical or any other extenuating condition or circumstance that may, in the opinion of the investigator and/or Amicus, pose an undue safety risk to the patient.
3. Concomitant use of miglitol (eg, Glyset), non-AT2221 form of miglustat (eg, Zavesca), acarbose (eg, Precose or Glucobay), voglibose (eg, Volix, Vocarb,or Volibo)

Ages: 0 Years to 17 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - UF Health Shands Hospital, Gainesville, Florida
- University Hospital of Padova, Padua, Italy
- National Taiwan University Hospital, Taipei, Taiwan